CLINICAL TRIAL: NCT05856526
Title: EvasayilTM : A Placebo-controlled Trial to Evaluate the Efficacy and Safety of Spesolimab in the Treatment of Patients With Netherton Syndrome
Brief Title: A Study to Test Whether Spesolimab Helps People With a Skin Disease Called Netherton Syndrome
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1368-0104; 2022-501104-10-00 (Registry Identifier: CTIS (EU)); U1111-1289-6825 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2023-04-26; First posted 2023-05-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Netherton Syndrome
MeSH Terms: conditions — Netherton Syndrome | interventions — spesolimab; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Spesolimab - solution for infusion; Drug: Placebo matching to spesolimab - solution for infusion; Drug: Spesolimab - solution for injection; Drug: Placebo matching to spesolimab - solution for injection
- Spesolimab (Experimental)
  Interventions: Drug: Spesolimab - solution for infusion; Drug: Placebo matching to spesolimab - solution for infusion; Drug: Spesolimab - solution for injection

INTERVENTIONS:
Drug: Spesolimab - solution for infusion — Solution for infusion
  Other Names: BI 655130
Drug: Placebo matching to spesolimab - solution for infusion — Solution for infusion
Drug: Spesolimab - solution for injection — Solution for injection
  Other Names: BI 655130
Drug: Placebo matching to spesolimab - solution for injection — Solution for injection
  Arms: Placebo

SUMMARY:
This study is open to people with a skin disease called Netherton syndrome (NS). People can join the study if they are 12 years or older. The purpose of this study is to find out whether a medicine called spesolimab helps people with NS.

Participants are divided into a spesolimab and a placebo group. Placebo injections look like spesolimab injections but do not contain any medicine. Every participant has a 2 in 3 chance of being in the spesolimab group. In the beginning, participants get the study medicine as an injection into a vein. Afterwards, they get it as an injection under the skin every month.

After 4 months, participants in the placebo group switch to spesolimab treatment.

Participants are in the study for up to 3 years. During this time, they visit the study site up to 42 times. The doctors regularly check participants' NS symptoms. The results are compared between the groups to see whether spesolimab works. The doctors also regularly check participants' general health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged 12 years and older (weight minimum is 35kg).
* Confirmed diagnosis of Netherton syndrome (NS) (causative SPINK5 mutations) at baseline (Visit 2).
* At least moderate severity of erythema at baseline (visit 2) (Ichthyosis Area Severity Index (IASI) score ≥ 16 and IASI-Erythema (E) score ≥8) and ≥ 3 on Investigator Global Assessment (IGA) score.
* Signed and dated written informed consent and assent in accordance with International Council on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission in the trial
* Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the clinical trial protocol (CTP) as well as in the patient, parent(s) (or patient's legal guardian) information.

Exclusion Criteria:

* Patients who have used topical corticosteroids (medium to high, US class I-V), topical retinoids, topical calcineurin inhibitors or keratolytics within 1 week prior to randomisation
* Patients who have used emollient on the area to be biopsied in the previous 24 hours
* Patients who have used systemic retinoids, other systemic immunosuppressants, systemic corticosteroids or phototherapy within 4 weeks prior to randomisation
* Patients who have used systemic antibiotics within 2 weeks prior to randomisation
* Patients who have received live vaccines within 4 weeks prior to randomisation
* Patients who have received investigational products, biologics or immunoglobulins within 4 weeks or 5 half-lives (whichever is longer) prior to randomisation
* Severe, progressive, or uncontrolled hepatic disease, defined as >3-fold Upper Limit of Normal (ULN) elevation in Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) or alkaline phosphatase, or >2-fold ULN elevation in total bilirubin
* Patients who have any prior exposure to BI 655130 or another interleukin 36 receptor (IL-36R) inhibitor biologics
* Further exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
IASI response | At baseline and at Week 16.
  Ichthyosis Area Severity Index (IASI) response is defined as a decrease of at least 50 % absolute change in IASI score from baseline at Week 16.

SECONDARY OUTCOMES:
Key secondary endpoint: IGA response | at Week 16.
  Investigator Global Assessment (IGA)
IGA score of 0 or 1 | up to Week 16.
  Investigator Global Assessment (IGA)
IASI response | At baseline and up to Week 12.
  Ichthyosis Area Severity Index (IASI)
IASI-E subscore response | At baseline and up to Week 16.
  Ichthyosis Area Severity Index - Erythema (IASI-E)
IASI-S subscore response | At baseline and up to Week 16
  Ichthyosis Area Severity Index - Scaling (IASI-S)
Percent change from baseline in IASI score | At baseline and up to Week 16.
  Ichthyosis Area Severity Index (IASI)
Absolute change from baseline in NRS pain | At baseline and up to Week 16.
  The Numeric Pain Rating Scale (NRS)
Absolute change from baseline in NRS itch | At baseline and up to Week 16.
  The Numeric Rating Scale (NRS)
Absolute change from baseline in DLQI score | At baseline and up to Week 16.
  Dermatology Life Quality Index (DLQI)
Absolute change from baseline in CDLQI score | At baseline and up to Week 16.
  Children Dermatology Life Quality Index (CDLQI)
The occurrence of treatment emergent adverse events including serious and/or opportunistic infections | up to 172 weeks.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (4):
  - Mission Dermatology Center, Rancho Santa Margarita, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Westmead Hospital, Westmead, New South Wales, Australia
- ASMC-IPSMC-skin and Veneral Diseases, Sofia, Bulgaria
- China (7):
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Southern Medical University Dermatology Hospital, Guangzhou
  - The Children's Hospital Zhejiang University School Of Medicine, Hangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Dermatology Hospital, Chinese Academy of Medical Sciences, Nanjing
  - Shanghai Skin Disease Hospital, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University, Shanghai
- HOP Saint-Louis, Paris, France
- Germany (3):
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Klinikum der Universität München AÖR, München
- Sourasky Medical Center, Tel Aviv, Israel
- Italy (2):
  - Istituto Dermopatico Dell'Immacolata - IDI - IRCCS, Roma
  - AO Città della Salute e Scienza, Torino
- Japan (3):
  - Nagoya University Hospital, Aichi, Nagoya
  - Juntendo University Urayasu Hospital, Chiba, Urayasu
  - Okayama University Hospital, Okayama, Okayama
- Hospital Tunku Azizah, Kuala Lumpur, Malaysia
- Erasmus MC - Sophia Kinderziekenhuis, Rotterdam, Netherlands
- ULS de São José, E.P.E. - Hospital Sto. António Capuchos, Lisbon, Portugal
- University Children Hospital Zürich, Zurich, Switzerland
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com
- See also: Related Info — https://www.firstskinfoundation.org/netherton-study-bi
- See also: Related Info — https://www.firstskinfoundation.org/userAssets/file/33023532_EVASAYIL_NS_Patient_info_sheet_US.pdf